CLINICAL TRIAL: NCT05987020
Title: Effects of Aromatherapy on Sleep Quality and Quality of Life for Older Adults at Risk of Metabolic Syndrome in the Community
Brief Title: Effects of Aromatherapy for Older Adults at Risk of Metabolic Syndrome in the Community
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: National Taipei University of Nursing and Health Sciences (Other)
Responsible Party: Principal Investigator, Mei-Hui Wang, Head nurse, National Taipei University of Nursing and Health Sciences
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: Mei-Hui Wang
Record Dates: First submitted 2023-07-27; First posted 2023-08-14 (Actual); Last update posted 2023-11-09 (Actual); Status verified 2023-11

CONDITIONS: Metabolic Syndrome
Keywords: Aromatherapy; Older Adults at Risk of metabolic syndrome; quality of life; quality of sleep
MeSH Terms: conditions — Metabolic Syndrome; Sleep Initiation and Maintenance Disorders | interventions — Aromatherapy

STUDY DESIGN:
Intervention Model Description: randomized controlled trial，RCT
Who Masked: Participant
Masking Description: single blinding
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- pre-specified group (Experimental): The experimental group received "aromatherapy", an intervention using lavender essential oil compound, while the control group received a placebo, sweet almond oil. The research tools include: "Basic Demographic Information", " The Chinese version of the Pittsburgh Sleep Quality Index, CPSQI ", "The World Health Organization Quality of Life Questionnaire -Taiwan Version" and ""The World Health Organization Quality of Life Questionnaire -old".
  Interventions: Other: Aromatherapy
- subgroup of participant (Placebo Comparator): The control group received a placebo, sweet almond oil. The research tools include: "Basic Demographic Information", " The Chinese version of the Pittsburgh Sleep Quality Index, CPSQI ", "The World Health Organization Quality of Life Questionnaire -Taiwan Version" and ""The World Health Organization Quality of Life Questionnaire -old".
  Interventions: Other: Aromatherapy

INTERVENTIONS:
Other: Aromatherapy — The experimental group received "aromatherapy", an intervention using lavender essential oil compound, while the control group received a placebo, sweet almond oil.

SUMMARY:
Background: According to statistics, Taiwan will become a super-aged society in 2025, and health promotion and care for the elderly are important issues of public health. With the prolongation of life, the older adults need to face their physical weakness, decline in psychological, cognitive and social related functional abilities, the prevalence of chronic diseases and the increase in the disabled population, which has a considerable impact on individuals, families and the overall social economy. However, most older adults suffering from chronic diseases are often accompanied by physical dysfunction, which affects the quality of sleep, causes emotional distress and emotional disorders, and leads to a decline in the quality of life. Studies have found that aromatherapy can not only improve sleep and emotional problems, but also relieve physical discomfort caused by diseases, achieve the purpose of reducing medical costs and improving quality of life. However, there are very few studies regrading older adults who are at risk of metabolic syndrome in community and the effects of inhalation of compound essential oils on their sleep and quality of life. Therefore, this study will explore the use of aromatherapy to improve the quality of sleep and life of the elderly. The research results can be used as a reference for community bases to promote the improvement of sleep and quality of life for older adults, so as to achieve the goal of healthy aging.

DETAILED DESCRIPTION:
Objective: The purpose of this study is to understand the sleep status and quality of life of the older adults at risk of metabolic syndrome in the community and the potential contributing factors, and to explore the effect of aromatherapy on improving the sleep quality and quality of life of the older adults at risk of metabolic syndrome in the community.

Methods: This study is a longitudinal study with a prospective randomized control design. A total of 64 elderly people were recruited from 2 community bases in the East District of Hsinchu City. The two bases were determined as the experimental group or the control group by simple randomization. The experimental group received "aromatherapy", an intervention using lavender essential oil compound, while the control group received a placebo, sweet almond oil. The research tools include: "Basic Demographic Information", " The Chinese version of the Pittsburgh Sleep Quality Index, CPSQI ", "The World Health Organization Quality of Life Questionnaire -Taiwan Version" and ""The World Health Organization Quality of Life Questionnaire -old".

Expected results: Older Adults in the experimental group (use aromatherapy) had better sleep and quality of life than those who use placebo.

ELIGIBILITY:
Inclusion Criteria:

Students aged 65 or above in community care bases 2. People with normal sense of smell 3. No severe respiratory disease 4. Have any one of the metabolic syndrome risk factors

According to the definition of the National Health Service:

1. Abdominal obesity: waist circumference ≧90cm for men, waist circumference ≧80cm for women;
2. High blood pressure: systolic blood pressure ≧ 130mmHg or diastolic blood pressure ≧ 85mmHg, or taking medication for hypertension prescribed by a doctor;
3. High fasting blood sugar: fasting blood sugar ≧100mg/dL, or taking a doctor's prescription for diabetes treatment;
4. High fasting triglycerides: ≧150mg/dL, or taking medicines for lowering triglycerides prescribed by doctors;
5. Low high-density lipoprotein cholesterol: men <40mg/dL, women <50mg/dL, the above five items are risk factors, and three or more items are met as metabolic syndrome.

5. Complaints of sleep disorders 6. Those who agree and can cooperate with research activities

Exclusion Criteria:

1. Those who are allergic to essential oils
2. Diagnosed with dementia, mental illness: such as depression
3. Cancer patients
4. Those who are currently using aromatherapy/have participated in or used aromatherapy-related activities within one month
5. Currently there is a wound on the shoulder and neck

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 64 (Estimated)
Dates: Start 2023-09-19 (Actual); Primary Completion 2023-11-08 (Actual); Study Completion 2024-04-30 (Estimated)

PRIMARY OUTCOMES:
The quality of sleep of elderly people at risk of metabolic syndrome in community bases participating in aromatherapy | 1 month after intervention
  Basic Demographic Information", " The Chinese version of the Pittsburgh Sleep Quality Index, CPSQI
The quality of life of elderly people at risk of metabolic syndrome in community bases participating in aromatherapy | 1 month after intervention
  Basic Demographic Information","The World Health Organization Quality of Life Questionnaire -Taiwan Version" and ""The World Health Organization Quality of Life Questionnaire -old".

CONTACTS AND LOCATIONS:
Locations (1):
- Hsinchu Cathay General Hospital, Hsinchu, East Dist, Taiwan

IPD SHARING:
Plan to Share IPD: No